CLINICAL TRIAL: NCT03747692
Title: Cairo University Faculty of Medicine
Brief Title: Intracervical Anasthesia in Outpatient Hystroscopy, Can Procedure be Completed Diagnostic and Therapeutic With no Need to General Anaesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Olfat Nooh Riad Ali, professor in cairo univerity, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: i18002
Record Dates: First submitted 2018-08-14; First posted 2018-11-20 (Actual); Last update posted 2018-11-20 (Actual); Status verified 2018-11

CONDITIONS: Infertility, Female
Keywords: intracervical anasthesia , outpatient hystroscopy ,
MeSH Terms: conditions — Infertility, Female | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: two groups will be used , 1st study group using intracervical anasthesia of a local anasthetic as Carbocaine3%,and 2nd group using NSAIDs and intracervical injection of a placebo ( saline ).Ask the patient to tell about any sense of nausea or vomiting or drowsiness.
Who Masked: Participant
Masking Description: group 1 will be subjected to intracervical injection of mepicaine hydrochloride 3%iof a local anasthetic as Carbocaine3% and group 2 will be subjected to intracervical injection of 5 ml of normal saline
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): patient put in dorsal postion , insertion of a speculum , sterilization of the cervix then intracervical injection of 5 ml mepicaine hydrochloride a local anasthetic as Carbocaine3%54 mg at site 3 and 9 using a 10 cm syringe
  Interventions: Procedure: study group
- control group (Placebo Comparator): patient receives one tablet of NSAIDs (diclofenac sodium 50 mg )15 minutes before procedure then 5 ml of normal saline will be injected intracervical using 10 cm syringe then wait for 5 minutes before the procedure
  Interventions: Procedure: control group

INTERVENTIONS:
Procedure: study group — local anesthesia by mepicaine hydrochloride by intracervical local injection using 10 mm syringe.
  Arms: study group
Procedure: control group — each patient receives one tablet of NSAIDs (diclofenac sodium 50 mg) and 5ml of a placebo in form of normal saline are injected intracervical 5 minutes before the procedure using 10 mm syringe.
  Arms: control group

SUMMARY:
Single blind randomized controlled study in which 80 patients coming for hystroscopy due to multiple indication as infertility, AUB and missed IUD were assigned for our study. Both Sample size and randomization were done by a computer program. Patients were classified into 2 groups, group 1 study group was subjected to intracervical injection of 5 mi of mepivacaine hydrochloride at position 3 and 9 of the vaginal portion of the cervix, and at least 5 minutes post injection before procedure done. The control group received NSAI injection 15 minutes before procedure and 5 ml of saline was injected in each side of cervix at 3 9 positions. Hystroscopy was done if an abnormality is detected an intervention was done. A descriptive scale of pain was done into mild, moderate or severe (that lead to interruption of the procedures).

DETAILED DESCRIPTION:
Procedures:

All patients were subjected to:

1. History taking
2. Verbal consent to participate in our study
3. Patient put in lithotomy position
4. Casco speculum was applied exposing the cervix
5. Betadine sterilization of the cervix then properly washed with saline as heavy metals of disinfectant may cause irritation with injection
6. Multiple toothed volselum was used just to fix cervix
7. 3 cartridges of mepivacaine hydrochloride was filled in 10 mi syringe
8. Do aspiration to exclude and avoid intravascular injection then infilterate slowly intracervical at both 3 and 9 positions
9. Instruments are removed and at least 5 minutes later procedure started.
10. Hystroscopy (rigid , 2.9 mm sheath) was introduced gently throw vaginoscopy exploring vagina , cervix and uterine cavity
11. Patient was monitored for pain all through the procedure by descriptive scale, mild, moderate and severe. ( moderate who needed to take rest then continue , severe that necessitated interruption of the procedure
12. All patients were monitored for signs of vaso vagal attack as sings (low blood pressure and bradycardia) before and if needed during. Occurrence of symptoms as pallor , sweet and fainting
13. All patients were monitored post procedure for persistence of colicky pain

ELIGIBILITY:
Inclusion Criteria:

1. must be under 40 years
2. must be no history of renal or hepatic disease
3. must be no known hypersensitivity to local anaesthetic agents
4. must be no significant vaginal or cervical infection.

Exclusion Criteria:

* All patients with history of sever vasovagal attack during any gynecological procedures.

Max Age: 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 80 (Actual)
Dates: Start 2018-08-15 (Actual); Primary Completion 2018-10-20 (Actual); Study Completion 2018-10-30 (Actual)

PRIMARY OUTCOMES:
tolerated hystroscopy | 30 minutes
  complete hystroscopy procedure with tolerable degree of pain.

SECONDARY OUTCOMES:
occurrence of complication | 30 minutes
  symptoms of vasovagal as vomiting , sweeting and bradycardia

CONTACTS AND LOCATIONS:
Locations (1):
- Outpatient Hystroscopy of Kasr El Ainy, Giza, Egypt